**Date:** March 30, 2018

**Official Title:** Preoperative and postoperative spatiotemporal gait parameters and gait asymmetry in patients with lumbar disc herniation: a prospective, cross-sectional study

## **Statistical Analysis Plan:**

The Statistical Package for Social Sciences (SPSS) version 23.0, was used for the all statistical analysis (SPSS Inc., Chicago, IL, USA). Normality was analyzed using the Kolmogorov Smirnov test. The Independent t-tests for parametric, or Mann-Whitney U tests for non-parametric data, was used to compare the means between the two groups for demographic characteristics, and all the spatiotemporal gait parameters. Also, kruskal-wallis test, were applied to determine differences between LDH levels groups for pain intensity. The Paired t-test and Wilcoxon test were used to analyze the spatiotemporal gait values and gait symmetry in the patients with LDH before and 15 days after surgery and between healthy controls and 15 days after surgery. A p-value of <0.05 was considered to indicate a statistically significant difference.